CLINICAL TRIAL: NCT01446653
Title: Reducing Alcohol Exposed Pregnancy Risk
Brief Title: Reducing Alcohol Exposed Pregnancy Risk: EARLY Randomized Controlled Trial
Acronym: EARLY RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, Associate Professor of Psychiatry and Neurobehavioral Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12794; R01AA014356 (NIH)
Record Dates: First submitted 2011-10-02; First posted 2011-10-05 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Exposed Pregnancy
Keywords: Fetal Alcohol Spectrum Disorders; FASDs; AEP risk; binge drinking; ineffective contraception
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Binge Drinking | interventions — Motivational Interviewing; Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EARLY (Experimental): Motivational Interviewing plus feedback counseling with information via video and brochures
  Interventions: Behavioral: Motivational Interviewing plus feedback
- Video Information (Active Comparator): Providing FASD information via documentary video clips
  Interventions: Behavioral: Video
- Informational Brochure (Active Comparator): Participants will receive informational brochures on contraception, women and drinking, and cutting down your drinking.
  Interventions: Behavioral: Informational Brochure

INTERVENTIONS:
Behavioral: Motivational Interviewing plus feedback — Provides an MI + feedback intervention supplemented with video and brochures-based information
  Arms: EARLY
Behavioral: Video — Video arm will provide information via documentary video
  Arms: Video Information
Behavioral: Informational Brochure — Informational Brochures are given to participants following baseline assessment.
  Arms: Informational Brochure

SUMMARY:
The EARLY Randomized Controlled Trial (RCT) will test the finalized EARLY preventive intervention against one comparison and one control condition. Because prevention of Alcohol-exposed pregnancy (AEP) will be achieved whether woman change drinking OR contraception, the primary endpoints will be rates of risky drinking and ineffective contraception at six-month follow-up, in addition to dichotomously defined "successful outcome" that will be observed whenever a woman has sufficiently altered one or both of the behaviors that placed her at risk of Alcohol-Exposed Pregnancy (AEP). The goal is to identify a transferable intervention that effectively reduces behaviors that put women at risk for AEP and alcohol-related birth defects including FASD.

DETAILED DESCRIPTION:
Drinking women are at risk for alcohol-exposed pregnancy (AEP) if they use contraception ineffectively. Binge drinking among women of childbearing age has increased, and risky frequent drinking has remained stable in this group of women. Although many women stop or reduce their drinking once they realize they are pregnant, pregnancy recognition does not occur until the 4th to 6th week of gestation for most women. Serious harm can occur to the fetus, especially between weeks 3 and 10 of gestation, if women drink during this period. Additionally, increasing numbers of women are drinking during pregnancy, despite public health warnings and scientific proof that alcohol is a teratogen. Although many women are aware of Fetal Alcohol Syndrome (FAS), few are aware that even low levels of alcohol exposure could lead to alcohol-related neurobehavioral disorders and alcohol-related birth defects (ARND, ARBD), now known as Fetal Alcohol Spectrum Disorders (FASD). Intervening before conception with women who are at risk for AEP could eliminate some cases of FASD. Women at risk are problem drinkers who fail to use contraception effectively, and those with ineffective contraception who sometimes drink at risk levels. Intervention could focus on postponing pregnancy among problem drinkers, or reducing drinking among women who forgo pregnancy prevention, or both.

Motivational interviewing focusing on the dual behaviors that compose risk for AEP is a promising approach. A five session, dual-focused motivational interviewing plus contraception counseling intervention was effective for women at risk for AEP who were not seeking treatment. Unfortunately, even though such interventions may prove effective, they are unlikely to be adopted in community settings due to their length and cost. What is needed is a less costly, transportable brief intervention that uses the effective components of these longer interventions, but delivers them in a condensed format. A briefer intervention could be used with women awaiting services or added to existing therapeutic services, and thus could have a larger public health impact on reducing the risk of AEP for women drawn from diverse settings. A single-session intervention, Project Balance, has shown evidence of efficacy with college women, but will require adaptation for less educated community-based women with more severe drinking problems or less contraception use. The next step needed to advance this field is to develop and test a less time-intensive intervention that builds on effective and theory-based interventions, and to test that intervention in women drawn from higher risk settings.

The purpose of this Stage 1b project is to develop and test the efficacy of a brief, theory-based, behavioral intervention among a high-risk community sample of fertile women who are at particularly high risk for an alcohol-exposed pregnancy (AEP). Because prevention of AEP will be achieved whether woman change drinking OR contraception, the primary endpoints will be rates of risky drinking and ineffective contraception at six-month follow-up, in addition to dichotomously defined "successful outcome" that will be observed whenever a woman has sufficiently altered one or both of the behaviors that placed her at risk of AEP. The goal is to identify a transferable intervention that effectively reduces behaviors that put women at risk for AEP and alcohol-related birth defects including FASD. The specific aims are to:

1. Develop the "Exploring Alcohol and Contraception Risks that Limit You" (EARLY) intervention, refine training methods and materials, and train therapists to deliver the intervention accurately.
2. Develop measures of the internal validity and fidelity of the intervention, and establish their psychometric properties.
3. Test the efficacy of the EARLY intervention against a minimal intervention condition that controls for the effects of assessment, time, and attention. Efficacy to retain participants, reduce drinking, and increase contraception will be tested in a pilot randomized trial of women drawn from the target populations: settings serving problem drinkers (outpatient drug and alcohol treatment settings) or women with ineffective contraceptive habits (STD and public health clinics)
4. Develop materials needed for a Stage 2 efficacy trial, including evidence of the feasibility and promise of the EARLY intervention, treatment manuals, therapist training materials, and a final instrumentation package.
5. Examine the role of variables other than group assignment (alcohol problem severity, psychiatric co-morbidity, drug use/severity, trans-theoretical model variables (readiness, stages, and processes of change, self efficacy, and therapeutic alliance) to mediate or moderate response, and examine secondary outcomes of the intervention, such as changes in readiness.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-44
* fertile
* can provide informed consent
* had vaginal intercourse with a man in the past 3 months
* uses ineffective or no contraception
* speaks and reads English
* reports drinking more than seven standard drinks per week on average or more than one binge drinking episode (more than 3 standard drinks on one occasion) during the past 3 months
* if opioid dependent with recent use, is enrolled in opiate agonist treatment
* planning to remain available for the follow-up period

Exclusion Criteria:

* pregnancy
* cognitive disorders including mental retardation, dementia, or active -psychosis that could impair ability to understand the intervention material or give informed consent
* current Major Depressive Disorder that could diminish responsiveness to interventions focused on promoting change
* currently opioid dependent with active use and not engaged in opiate agonist treatment
* concurrently participating in another behavioral intervention study during the study period targeting drinking or contraception efficacy that could interfere with or augment the intervention in the EARLY project.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2007-02; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Drinks per drinking day | 6 months
Rate of effective contraception | 6 months

SECONDARY OUTCOMES:
Alcohol Exposed Pregnancy risk | 6 months
  Risk for AEP is defined as the proportion of women who no longer meet the entry criteria for the trial based on her use of alcohol and unprotected intercourse, measured via the TLFB. Specifically, this means that the woman is 1) no longer at risk for pregnancy due to perfect contraception or abstinence; and/or 2) is drinking at or below recommended levels (<8drinks per week with no binges).

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Ingersoll, Ph.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE, Richmond, Virginia

REFERENCES:
- [Result] Ingersoll KS, Hettema JE, Cropsey KL, Jackson JP. Preconception markers of dual risk for alcohol and smoking exposed pregnancy: tools for primary prevention. J Womens Health (Larchmt). 2011 Nov;20(11):1627-33. doi: 10.1089/jwh.2010.2633. Epub 2011 Aug 12. PMID 21838526
- [Result] Fabbri S, Farrell LV, Penberthy JK, Ceperich SD, Ingersoll KS. Toward prevention of alcohol exposed pregnancies: characteristics that relate to ineffective contraception and risky drinking. J Behav Med. 2009 Oct;32(5):443-52. doi: 10.1007/s10865-009-9215-6. Epub 2009 May 21. PMID 19459039
- [Result] Ingersoll KS, Ceperich SD, Hettema JE, Farrell-Carnahan L, Penberthy JK. Preconceptional motivational interviewing interventions to reduce alcohol-exposed pregnancy risk. J Subst Abuse Treat. 2013 Apr;44(4):407-16. doi: 10.1016/j.jsat.2012.10.001. Epub 2012 Nov 26. PMID 23192220
- [Result] Farrell-Carnahan L, Hettema J, Jackson J, Kamalanathan S, Ritterband LM, Ingersoll KS. Feasibility and promise of a remote-delivered preconception motivational interviewing intervention to reduce risk for alcohol-exposed pregnancy. Telemed J E Health. 2013 Aug;19(8):597-604. doi: 10.1089/tmj.2012.0247. Epub 2013 Jun 13. PMID 23763608
- [Result] Penberthy JK, Hook JN, Hettema J, Farrell-Carnahan L, Ingersoll K. Depressive symptoms moderate treatment response to brief intervention for prevention of alcohol exposed pregnancy. J Subst Abuse Treat. 2013 Oct;45(4):335-42. doi: 10.1016/j.jsat.2013.05.002. Epub 2013 Jun 28. PMID 23810264
- [Result] Hettema J, Cockrell S, Russo J, Corder-Mabe J, Yowell-Many A, Chisholm C, Ingersoll K. Missed Opportunities: Screening and Brief Intervention for Risky Alcohol Use in Women's Health Settings. J Womens Health (Larchmt). 2015 Aug;24(8):648-54. doi: 10.1089/jwh.2014.4961. Epub 2015 Jul 31. PMID 26230758